CLINICAL TRIAL: NCT00672763
Title: The Immunomodulatory Role of Vitamin D in Inflammatory Bowel Disease (The IBDVit Study): Double-Blind, Placebo-Controlled Trial of Adjuvant Vitamin D (Colecalciferol) With Corticosteroids in Active Crohn's Disease
Brief Title: Adjuvant Vitamin D With Corticosteroids in Active Crohn's Disease
Acronym: IBDVit1
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit adequate trial participants
Sponsor: Imperial College London (Other)
Responsible Party: Dr. Andrew N. Milestone, Imperial College London
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VITDIBD1; EudraCT: 2007-006692-37
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Inflammatory Bowel Disease; Vitamin D; Randomised; Placebo
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Calcium; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Standard corticosteroid treatment PLUS Vitamin D3 (Colecalciferol).
  Interventions: Drug: Colecalciferol D3 (Vigantol Oil)
- B (Placebo Comparator): Standard corticosteroid treatment PLUS placebo (Migliol Oil)
  Interventions: Drug: Medium chain triglycerides

INTERVENTIONS:
Drug: Colecalciferol D3 (Vigantol Oil) — 1. Standard oral Prednisolone 40mg daily (or Budesonide 9mg daily) for 4 weeks;
  2. Supplemental calcium and vitamin D3 (CalcichewD3Forte) 1000mg and 800iU respectively daily for duration of steroid treatment;
  3. Colecalciferol 100,000iU orally once fortnightly for 4 weeks (2 doses).
  Other Names: CalcichewD3Forte (Calcium and Vitamin D3); Vigantol Oil (Colecalciferol D3)
  Arms: A
Drug: Medium chain triglycerides — 1. Standard oral Prednisolone 40mg daily (or Budesonide 9mg daily) for 4 weeks;
  2. Supplemental calcium and vitamin D3 (CalcichewD3Forte) 1000mg and 800iU respectively daily for duration of steroid treatment;
  3. Migliol Oil 5ml oral fortnightly (2 doses)
  Other Names: CalcichewD3Forte (Calcium and Vitamin D3); Migliol Oil (Placebo)
  Arms: B

SUMMARY:
The purpose of this study is to determine whether the addition of vitamin D to standard corticosteroids improves onset of remission in active Crohn's Disease, a form of Inflammatory Bowel Disease (IBD).

DETAILED DESCRIPTION:
Crohn's Disease is a form of Inflammatory Bowel Disease (IBD). It is caused by abnormal immune-mediated gut inflammation and is both chronic and difficult to treat. Symptoms are often unpleasant (e.g. abdominal pain, diarrhoea, disfiguring fistulation) and often lead to surgery to remove diseased bowel.

There is emerging evidence that Vitamin D, a nutrient largely produced in the skin upon exposure to sun-light, may possess properties regulating the immune system in IBD. In addition, vitamin D deficiency appears common in Inflammatory Bowel Disease.

This study aims to determine if the addition of vitamin D to standard corticosteroid treatment in active Crohn's Disease helps to achieve remission (resolution of symptoms).

ELIGIBILITY:
Inclusion Criteria:

1. Active Crohn's Disease Activity (CDAI) Score >200 to 450;
2. Diagnosis of IBD and distribution of disease previously confirmed
3. The participant able to give informed consent form;
4. Stable doses of the following concurrent IBD medications prior to inclusion:

   * 5-aminosalicylates (≥4 weeks)
   * Thiopurines (≥8 weeks)
   * No corticosteroids (within 4 weeks)
   * No biological agents (within 8 weeks).

Exclusion Criteria:

1. Unable to give informed written consent;
2. Co-existence of any other chronic inflammatory conditions
3. Failure to meet concurrent IBD medication criteria;
4. Hypercalcaemia (Corrected serum calcium > 2.66 mmol/L) or history of vitamin D hypersensitivity;
5. Diagnosis of any of the flowing: active tuberculosis, sarcoidosis, hyperparathyroidism, pseudohyperparathyroidism, nephrolithiasis, silicosis, liver failure, renal failure or malignancy, active TB, sarcoidosis or lymphoma or other granulomatous disease;
6. Known intolerance or contraindication to vitamin D or trial medication (i.e. corticosteroids / infliximab);
7. Biochemical disturbance at enrolment: serum corrected calcium > 2.66 mmol/L) or serum creatinine >250 micromol/L;
8. Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Clinical Remission (CDAI score <150) | 4 Weeks

SECONDARY OUTCOMES:
Reduction in CDAI suggestive of a clinical improvement. | Week 4
Reduction in serum C-reactive protein. | Week 4
Reduction of faecal calprotectin levels | Week 4
Clinical Remission (CDAI score <150) | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Andrew N Milestone, BSc(Hons) MBBS MRCP, Principal Investigator — Imperial College London (Hammersmith and St. Mark's Hospitals); Subrata Ghosh, MD (Edin) FRCP, FRCP (Edin), Study Chair — Imperial College London (Hammersmith Hospital); Ailsa L Hart, BA(Hons), BM BCh, MRCP, PhD, Study Director — Imperial College London (St. Mark's Hospital)
Locations (2):
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust (Hammersmith, Charing Cross and St. Mary's Hospitals), London, London
  - St. Mark's Hospital, Harrow, Middlesex